CLINICAL TRIAL: NCT07062809
Title: Comparative Effects of Sub-Occipital Myofascial Release With and Without Sustained Natural Apophyseal Glide Among Patients With Cervicogenic Dizziness.
Brief Title: Comparing the Effects of Sub-Occipital Myofascial Release With and Without SNAG on People With Cervicogenic Dizziness.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0170
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Dizziness; Cervicogenic Headache
Keywords: Cervicogenic Dizziness; Pain; Suboccipital Myofascial Release
MeSH Terms: conditions — Dizziness; Post-Traumatic Headache; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub Occipital Myofascial release and Sustained Natural Apophyseal Glide (SNAGS). (Active Comparator): The patient will instruct to be seated then will turned his head toward direction that will cause his dizziness. when subject will turn his head, The manual therapist will perform a constant PA glide (using his thumbs one over the other) to upper cervical C1 or C2 vertebra (Oriented toward patient's eyeballs). If flexion or extension movement will provoke the dizziness, an anterior glide will apply to the C2 spinous process. If rotation will provoke dizziness, then an anterior glide will be applied to the C1 transverse process. The patient will be free from the symptoms and will be instructed to discontinue movement when somewhat vertigo happened through the glide Implementation. In the beginning treatment period, that procedure will repeat six times. During the following therapy , Mulligan SNAGs will perform ten repetitions and mild excess compression will be used only if no vertigo will feel.
  Interventions: Other: Sub Occipital Myofascial release and (SNAGS).
- Sub Occipital Myofascial release (Active Comparator): When using the technique, the patient will be in Upward-facing position with their head fully aided on the therapist's hands. The therapist will put three middle fingers simply inferior to the nuchal line, raise the tips of the fingers in the direction of the ceiling, and then simply pull them upward. This process will be performed three times a week on different days for two to three minutes, with five to seven times.
  Interventions: Other: Sub Occipital Myofascial release.

INTERVENTIONS:
Other: Sub Occipital Myofascial release and (SNAGS). — The patient will instruct to be seated then will turned his head toward direction that will cause his dizziness. when subject will turn his head, The manual therapist will perform a constant PA glide (using his thumbs one over the other) to upper cervical C1 or C2 vertebra (Oriented toward patient's eyeballs). If flexion or extension movement will provoke the dizziness, an anterior glide will apply to the C2 spinous process. If rotation will provoke dizziness, then an anterior glide will be applied to the C1 transverse process.
  Arms: Sub Occipital Myofascial release and Sustained Natural Apophyseal Glide (SNAGS).
Other: Sub Occipital Myofascial release. — When using the technique, the patient will be in Upward-facing position with their head fully aided on the therapist's hands. The therapist will put three middle fingers simply inferior to the nuchal line, raise the tips of the fingers in the direction of the ceiling, and then simply pull them upward.
  Arms: Sub Occipital Myofascial release

SUMMARY:
Cervicogenic dizziness is defined as a sensation of rotation, resulting from an alteration of the neck proprioceptive afferents of the upper cervical spine.Sub-occipital Release, a type of Myofascial Release (MFR) is a form of manual therapy technique which can be used for the treatment of cervicogenic dizziness. Sub-occipital muscles, dura matter and C2 vertebrae are connected to each other through the fascia. Sustained natural apophyseal glides (SNAGs) are also an effective treatment for cervicogenic dizziness. This study aim to determine Comparative Effect of Sub-Occipital Myofascial release with and without Sustained Natural Apophyseal Glide among patients with Cervicogenic Dizziness.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted in Hameed Latif Teaching Hospital and National hospital & Medical Center. Non-probability consecutive sampling will be used to collect the data. Subjects with age group between 22 to 54 years old will be taken. Data will be collected from the patients having present complaint of cervicogenic dizziness. Group A and Group B were the two randomly selected groups into which the participants were divided. Baseline assessment of pain, dizziness and Headache was taken using Visual Analogue Scale (VAS), Dizziness Handicap Inventory (DHI) and Numeric Pain Rate Scale (NPRS) respectively, before the start of treatment by an assessor. Subjects will be selected on the basis of inclusion and exclusion criteria. Both the Groups will receive Hot Pack ,TENS , Ultrasound ,and also will receive Sternocleidomastoid, Trapezius, Scalene, and Pectoralis minor muscle stretching exercises, while Group A will receive Sub-Occipital Myofascial Release and Sustained Natural Apophyseal Glide (SNAG), and Group B will receive Sub Occipital Myofascial Release. Short term effects would be assessed after treatment for 3 sessions per week on alternate days for 4 weeks. Data analysis will be done by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Cervicogenic dizziness patients both male and female.
* Age group between 22 to 54 Years old.
* Passive Accessory Assessment of the UCS (C0-1, C1-2, C2-3).
* Dizziness related to either movements or positions of the cervical spine, or occurring with a stiff or painful neck.
* Symptoms > 3 months.
* Moderate disability score on the Dizziness Handicap Inventory (DHI) [31-60 points] .

Exclusion Criteria:

* Conditions for which manual therapy is contraindicated
* Traumatic brain injury
* Previous surgery to the upper cervical spine and marked cervical spine disc protrusion
* By neurologist .Vestibular disorders (e.g. Benign Paroxysmal Positional Vertigo, Meniere's disease, peripheral vestibulopathy)

  * CNS disorder (e.g.cerebellar ataxia, stroke, demyelination)
  * Migraine associated vertigo
  * Psychogenic dizziness
  * Cardiovascular disorders

Ages: 22 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 4 weeks
  The dizziness intensity was registered with a VAS, a valid and reliable tool for measuring dizziness intensity (reliability test-retest of this VAS is r = 0.85-0.96) .A continuous vertical line of 100 mm was anchored by two verbal descriptors ("no dizziness" and "worst imaginable dizziness"), and each end of the line had a mark; the subjects had to mark on the line the worst perceived dizziness since the last appointment (wVAS). Although it is a subjective and individual scale of the patient, it allows us to register the intensity of dizziness quickly, and its use in the clinic is widespread.

SECONDARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | 4 weeks
  The impact of dizziness on quality of life is often assessed by the Dizziness Handicap Inventory (DHI). The DHI contains 25 items, and a total score (0-100 points) is obtained by summing ordinal scale responses, higher scores indicating more severe handicap. The scale was developed to capture various sub-domains of self-perceived handicap and comprises 7 physical, 9 functional, and 9 emotional questions

OTHER OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 4 weeks
  This scale will be used to measure the patient's level of pain. The numbers on this scale go from 0 to 10. "No pain" is denoted by a score of 0, and "worst pain" by a score of 10. High test-retest reliability has been demonstrated using NPRS (r = 0.96 and 0.95, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Muzna Munir, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Hameed Latif Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoppes CW, Romanello AJ, Gaudette KE, Herron WK, McCarthy AE, McHale CJ, Bares J, Turner R, Whitney SL. Physical therapy interventions for cervicogenic dizziness in a military-aged population: protocol for a systematic review. Syst Rev. 2020 Mar 23;9(1):62. doi: 10.1186/s13643-020-01335-4. PMID 32293544
- [Background] Yaseen K, Hendrick P, Ismail A, Felemban M, Alshehri MA. The effectiveness of manual therapy in treating cervicogenic dizziness: a systematic review. J Phys Ther Sci. 2018 Jan;30(1):96-102. doi: 10.1589/jpts.30.96. Epub 2018 Jan 27. PMID 29410575
- [Background] Chu EC, Zoubi FA, Yang J. Cervicogenic Dizziness Associated With Craniocervical Instability: A Case Report. J Med Cases. 2021 Nov;12(11):451-454. doi: 10.14740/jmc3792. Epub 2021 Nov 5. PMID 34804305
- [Background] De Vestel C, Vereeck L, Van Rompaey V, Reid SA, De Hertogh W. Clinical characteristics and diagnostic aspects of cervicogenic dizziness in patients with chronic dizziness: A cross-sectional study. Musculoskelet Sci Pract. 2022 Aug;60:102559. doi: 10.1016/j.msksp.2022.102559. Epub 2022 Mar 26. PMID 35364427
- [Background] Sung YH. Suboccipital Muscles, Forward Head Posture, and Cervicogenic Dizziness. Medicina (Kaunas). 2022 Dec 5;58(12):1791. doi: 10.3390/medicina58121791. PMID 36556992
- [Background] Kuculmez O, Coban K, Sukun A. Prevalence of cervicogenic dizziness in patients with neck pain and effectiveness of cervicogenic dizziness rehabilitation. 2024.
- [Background] Gill-Lussier J, Saliba I, Barthelemy D. Proprioceptive Cervicogenic Dizziness Care Trajectories in Patient Subpopulations: A Scoping Review. J Clin Med. 2023 Feb 27;12(5):1884. doi: 10.3390/jcm12051884. PMID 36902670
- [Background] Reid SA, Callister R, Snodgrass SJ, Katekar MG, Rivett DA. Manual therapy for cervicogenic dizziness: Long-term outcomes of a randomised trial. Man Ther. 2015 Feb;20(1):148-56. doi: 10.1016/j.math.2014.08.003. Epub 2014 Aug 27. PMID 25220110
- [Background] Reid SA, Rivett DA, Katekar MG, Callister R. Comparison of mulligan sustained natural apophyseal glides and maitland mobilizations for treatment of cervicogenic dizziness: a randomized controlled trial. Phys Ther. 2014 Apr;94(4):466-76. doi: 10.2522/ptj.20120483. Epub 2013 Dec 12. PMID 24336477
- [Background] Carrasco-Uribarren A, Pardos-Aguilella P, Perez-Guillen S, Lopez-de-Celis C, Rodriguez-Sanz J, Cabanillas-Barea S. Combination of Two Manipulative Techniques for the Treatment of Cervicogenic Dizziness: A Randomized Controlled Trial. Life (Basel). 2022 Jul 9;12(7):1023. doi: 10.3390/life12071023. PMID 35888111